CLINICAL TRIAL: NCT01774383
Title: Investigating the Pathophysiological Roles of Cortical, Sub-thalamic Nuclear and Pedunculo-pontine Nuclear Oscillation in Movement Termination of Parkinson Disease Patients
Status: Completed | Type: Observational
Sponsor: China Medical University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Principal Investigator, Chon-Haw Tsai, The Chief, Department of Neurology, China Medical University Hospital
Other Study IDs: DMR101-IRB2-005
Record Dates: First submitted 2013-01-21; First posted 2013-01-24 (Estimated); Last update posted 2014-01-30 (Estimated); Status verified 2014-01

CONDITIONS: Parkinson's Disease; Deep Brain Stimulation
Keywords: Parkinson's disease; sub-thalamic nucleus; oscillation; local field potential
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The ERD and ERS patterns of coordination between the STN and cortical regions in the termination of volitional movement in PD patients.

DETAILED DESCRIPTION:
The project will investigate the roles of cortical regions, sub-thalamic nucleus and pedunculo-pontine nucleus in the preparation of volitional movement termination in patients with Parkinson's disease (PD)receiving deep brain stimulation. Currently there are two models of inhibitory preparation of volitional movements. The "withdrawal mechanism" posits the explanation that movement termination is due to the"shutting off" of the activated neuralcircuitry, whereas the "inhibition mechanism" suggests that inhibitory neural structures are activated to terminate the voluntary movement. These hypotheses were deduced from the study of scalp movement-related cortical potential recordings and how the deep structures involved in the execution in movement termination is uncertain. Movement preparation prior to movement onset (Mon) has been addressed in both scalp recordings of MRCP and from recent studies of STN in PD patients. However,the electro-physiologic information concerning the role of STN in the preparation of movement offset (Moff)is less understood. In our pilot study, we have found that high-beta event-related de-synchronization (ERD)appeared earlier (3 seconds prior to Mon) than those of low-beta and alpha for the Mon phasic movement.There was no alpha ERD for the Mon tonic movement. Alpha, low-beta, and high-beta ERD all appeared about 1 second prior to the Moff tonic movement. These findings suggest that STN participates in the preparation of volitional movement termination but via different mechanism from that in movement initiation.Unlike asynchronous ERD frequency bands present in movement initiation, a simultaneous ERD across wide frequency bands in STN may play a pivotal role in terminating volitional movement. Since there is tight connection between the cortical regions and STN, it is intriguing to know the relationship of these oscillatory patterns between the deep and superficial neural structures. In the current proposal, we will examine the patterns of ERD and ERS prior to Mon and Moff of tonic movements in both cortical and STN regions and determine the temporal relationship among them.

ELIGIBILITY:
Inclusion Criteria:

Patients with PD undergoing deep brain stimulation. The inclusion criteria for the patient selection will be those with motor complications (wearing off, on-off, drug-induced dyskinesia). Levodopa challenge test will be conducted to ensure good beneficial response of medication in each patient, since this is a reliable indicator to predict the DBS effect.

Exclusion Criteria:

1. impairment of cognition that leads unable to fully cooperate with the oral commands during operation,
2. any moderate to severe medical disorders such as poor control of diabetic mellitus, functional III or above congestive heart failure, or cancer with distant metastasis etc.,
3. severe mood disorders such as major depression.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PD undergoing deep brain stimulation of the sub-thalamic nucleus.
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2012-08; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
The ERD and ERS patterns of coordination between the STN and cortical regions in the termination of volitional movement in PD patients. | after deep brain stimulation 4th day
  1. To investigate the functional connectivity between the sub-thalamic nucleus and cerebral cortex on movement initiation and termination in PD patients.
  2. To examine phase leading roles of sub-thalamic nucleus and cerebral cortex in conducting volitional movements and will mainly focus on the movement termination.

CONTACTS AND LOCATIONS:
Overall Officials: Chon-Haw Tsai, MD, PHD, Principal Investigator — Department of Neurology, China Medical University Hospital, Taichung, Taiwan
Locations (1):
- China Medical University Hospital/Neuro Depart., Taichung, Taiwan, Taiwan